CLINICAL TRIAL: NCT00855426
Title: Diagnostic Protocol Of Painful Hip
Status: Suspended | Type: Observational
Why Stopped: the research is on susoension beacause the lack of manpower
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Ori Safran, Hadassah Medical Organization
Other Study IDs: SAF03-HMO-CTIL
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-10

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Nondisplaced hip fractures may be radiographically occult and require MRI or single photon emission CT bone scintigraphy for accurate diagnosis. Both examinations are expensive and are not readily available in many hospitals. Ultrasound (US) examination is relatively inexpensive and preliminary data had demonstrated its efficacy in detecting occult fractures in other sites. Our objective is to evaluate US examination as a screening tool for occult hip fractures in posttraumatic painful hips in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women above 40 years old
2. Trauma to the hip .
3. Extreme difficulty in walking or inability to step on the leg, following sensitivity in the hip joint area after local pressure or in a movement.
4. X ray of the pelvis aimed to the suspected hip joint (including AP lateral position and internal rotation) does not demonstrate fracture in the joint or the pelvis.

Exclusion Criteria:

1. None

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that are admitted to the ER after trauma.
Sampling Method: Non-Probability Sample